CLINICAL TRIAL: NCT00786578
Title: Evaluation of Intramyocellular Lipid Content (IMCL) in Skeletal Muscle by Magnetic Resonance Spectroscopy
Brief Title: Evaluation of Skeletal Muscle Lipid Content by Magnetic Resonance Spectroscopy
Status: Withdrawn | Type: Observational
Why Stopped: not funded
Sponsor: University of Minnesota (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0708M13941; 5K12RR023247-02 (NIH)
Record Dates: First submitted 2008-11-05; First posted 2008-11-06 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
Keywords: training; intramyocellular lipid; insulin resistance
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood will be sampled and retained for future metabolic testing as needed
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: overweight runners (BMI>25)
- 2: lean runners (BMI<24)

SUMMARY:
Type 2 diabetes is a growing public health issue and one component of Type 2 diabetes is 'insulin resistance" - the ability of insulin to work less well. The skeletal muscle is one of the largest users of sugar in the body, when the skeletal muscle is "insulin resistant", this contributes to diabetes. There is some evidence that the amount of fat in the skeletal muscle is related to the amount of insulin resistance. We are asking people to participate in a study to look at the amount of fat in muscle and how this fat amount changes with exercise. We hypothesize that heavier people will have higher amounts of fat and deplete this fat more slowly than lean subjects.

DETAILED DESCRIPTION:
High intramyocellular lipid (IMCL) content in skeletal muscle has been correlated to insulin resistance in obese subjects. Yet, endurance athletes have high intramyocellular lipid content and very low insulin resistance. There are several explanations for this paradox. This study will use a new magnetic resonance imaging technique to look at the amount of fat in the muscle and its depletion with exercise. We hypothesize that overweight subjects will have higher amounts of fat and deplete this fat more slowly than lean subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age range will be from age 18 to 45. We will be limiting the upper age range because increased age is associated with sarcopenia and alteration of fiber type.
* We will define the lean trained group by a BMI of < 24 kg/m2. We will define the overweight group as BMI > 26 25 kg/m2.
* The subjects should be participating in regular running exercise (> 30 min/day, ≥ 5 days/week).
* Weight must be stable [+/- 5 pounds] for at least the three months prior to the study for all participants.

Exclusion Criteria:

* The subjects must not be on medications that may affect lipid levels, specifically lipid lowering agents, birth control pills, or diuretics.
* The subjects should not be on a high fat diet (> 45% fat) as measured by a screening questionnaire.
* The subject must not have any contraindications to magnetic resonance imaging.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy subjects on regular running program.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
absolute change in intramyocellular lipid quantity with exercise | over 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Lisa S Chow, Principal Investigator — University of Minnesota
Locations (1):
- Univeresity of Minnesota, Minneapolis, Minnesota, United States